CLINICAL TRIAL: NCT03914378
Title: The Effects on Auditory Function of RADiotherapy and Chemotherapy Treatments for Head and Neck Tumours (EARAD)
Acronym: EARAD
Status: Recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Professor Chris Plack, Ellis Llwyd Jones Professor of Audiology, University of Manchester
Other Study IDs: NHS001435
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Neoplasms; Hearing Loss
Keywords: Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour blocks.
  One 10 ml (two teaspoons) blood sample at each time point:
  1. Baseline (2 repeats)- one repeat at the planning scan and one repeat on day 1 of RT (prior to RT)
  2. Further time points: one per week throughout treatment (5 time points)
  3. Final visit: one 10ml EDTA blood to be taken at 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Discovery Phase - Radiotherapy only: 25 patients undergoing radiotherapy only for head / neck cancer
- Discovery Phase - Radiotherapy plus chemotherapy: 25 patients undergoing radiotherapy plus chemotherapy for head / neck cancer
- Validation Phase - Radiotherapy only: 25 patients undergoing radiotherapy only for head / neck cancer
- Validation Phase - Radiotherapy plus chemotherapy: 25 patients undergoing radiotherapy plus chemotherapy for head / neck cancer
- Retrospective Cohort: 50 patients who previously received unilateral radiotherapy for head / neck cancer up to 5 years post-treatment
- Normal Hearing Controls for Retrospective Cohort: 50 controls with normal hearing, age- and sex-matched to retrospective cohort
- Hearing Impaired Controls for Retrospective Cohort: 50 controls with impaired hearing, age-, sex-, and audiogram-matched to retrospective cohort

SUMMARY:
Radiotherapy and combined radiotherapy and chemotherapy are used to treat most tumours in the head and neck region. Unfortunately, these treatments often result in hearing loss and tinnitus that has a negative impact on quality of life. This study will use a battery of sensitive tests, including measures of hair cell and neural function, before and after treatment, to measure the effects of these treatments on auditory function. The results will be compared with the individual radiotherapy dose characteristics, using state-of-the-art data mining technology, to identify the auditory substructures that are most sensitive to radiation with respect to the effects on auditory function. The data will provide the basis for new dose constraints to limit radiation doses to any identified substructures and to minimise loss in hearing ability for patients undergoing treatment for head and neck cancer.

DETAILED DESCRIPTION:
The overall aim is to provide the data that will define radiotherapy dose constraints for individual substructures of the auditory pathway such that a better balance can be made between hearing loss and tumour control during radiotherapy for head and neck cancer. In particular the study aims to:

1. Determine the impact of radiotherapy to the head and neck region on auditory function, including measures of hair cell and neural function
2. Determine the interaction between radiation and cisplatin chemotherapy on auditory function
3. Determine relations between different functional effects and radiation dose to substructures within the ear using advanced voxel-based data mining techniques
4. Determine the auditory substructure that is most associated with speech-in-noise deficits
5. Identify and validate a test which is most predictive of damage to that substructure, and could be the basis for future diagnosis
6. Validate the importance of the localised sensitive substructure in an independent cohort

ELIGIBILITY:
For Prospective Patient Cohorts:

Inclusion Criteria:

* Diagnosed with head and neck cancer
* An MDT treatment decision of radiotherapy +/- cisplatin based chemotherapy

Exclusion Criteria:

* Hearing loss greater than 25 dB HL (average from 0.25 to 4 kHz) prior to the study
* Existing hearing loss (self-reported- need for hearing aid)
* An MDT treatment decision of carboplatin based chemotherapy
* Involved in another research project where the treatment is known to be ototoxic
* Unable to give informed consent

For Retrospective Patient Cohort:

Inclusion Criteria:

* Previously diagnosed and treated for head and neck cancer
* Radiotherapy treatment to one side of the head
* Within 5 years post-treatment
* An MDT treatment decision of radiotherapy +/- cisplatin based chemotherapy

Exclusion Criteria:

* An MDT treatment decision of carboplatin based chemotherapy
* Unable to give informed consent

For Retrospective Normal-Hearing Controls:

Exclusion Criteria:

* Hearing loss greater than 20 dB HL (at any octave frequency from 0.25 to 4 kHz)
* Unable to give informed consent

For Retrospective Hearing-Impaired Controls:

Inclusion Criteria:

* Hearing loss greater than 20 dB HL (average from 0.25 to 4 kHz)

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer and controls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Audiology test results for prospective cohort | T1 =baseline, before radiotherapy and T2= 3 months following radiotherapy.
  For prospective patients undergoing radiotherapy to one side of the head, comparison of the test outcomes between the patient's two ears at baseline and 3 months, and relation to radiation dose characteristics.
  For prospective patients undergoing radiotherapy to both sides of the head, comparison of the test outcomes for both ears at baseline and at 3 months, and relation to radiation dose characteristics.
Audiology test results for retrospective cohort | A single timepoint within 4 years post-treatment
  Comparison of test outcomes between treatment and non-treatment ears and relation to radiation does characteristics. Further comparison with hearing impaired and normal hearing control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03914378/Prot_SAP_003.pdf